CLINICAL TRIAL: NCT02930694
Title: A Randomized, Open-label, 2-Way Crossover, Parallel-group Study in Healthy Male and Female Subjects to Evaluate the Bioavailability, Safety and Tolerability of a Solid Dosage Formulation Relative to a Suspension of JNJ-54175446
Brief Title: A Study to Evaluate the Bioavailability, Safety and Tolerability of a Solid Dosage Formulation Relative to a Suspension of JNJ-54175446 in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108246; 54175446EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-54175446; Capsules; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Treatment Sequence AB (Experimental): Participants will receive Treatment A [JNJ-54175446, 50 milligram (mg) capsule] on Day 1 of period 1 followed by Treatment B [JNJ-54175446, 50 mg suspension] on Day 1 of period 2. Both the treatment periods will be separated by washout period of minimum 10 days.
  Interventions: Drug: JNJ-54175446 (capsule); Drug: JNJ-54175446 (suspension)
- Group 1: Treatment Sequence BA (Experimental): Participants will receive Treatment B on Day 1 of period 1 followed by Treatment A on Day 1 of period 2. Both the treatment periods will be separated by washout period of minimum 10 days.
  Interventions: Drug: JNJ-54175446 (capsule); Drug: JNJ-54175446 (suspension)
- Group 2: Treatment Sequence CD (Experimental): Participants will receive Treatment C [JNJ-54175446, 100 mg capsule] on Day 1 of period 1 followed by Treatment D [JNJ-54175446, 100 mg suspension] on Day 1 of period 2. Both the treatment periods will be separated by washout period of minimum 10 days.
  Interventions: Drug: JNJ-54175446 (capsule); Drug: JNJ-54175446 (suspension)
- Group 2: Treatment Sequence DC (Experimental): Participants will receive Treatment D on Day 1 of period 1 followed by Treatment C on Day 1 of period 2. Both the treatment periods will be separated by washout period of minimum 10 days.
  Interventions: Drug: JNJ-54175446 (capsule); Drug: JNJ-54175446 (suspension)

INTERVENTIONS:
Drug: JNJ-54175446 (capsule) — Participants will receive JNJ-54175446 capsule at a dose of 50 mg or 100 mg, orally.
Drug: JNJ-54175446 (suspension) — Participants will receive JNJ-54175446 suspension at a dose of 50 mg or 100 mg, orally.

SUMMARY:
The primary purpose of the study is to investigate the plasma pharmacokinetics and bioavailability (BA) of a single dose of a solid dose formulation with 2 different strengths of JNJ-54175446 (50 milligram [mg] and 100 mg capsules) relative to the suspension of JNJ-54175446 under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) between 18 and 32 kilogram per square meter (kg/m^2), inclusive (BMI = weight/height^2)
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) [inclusive QTcF less than or equal to (<=) 450 millisecond (msec) for males and <= 470 msec for females] performed at screening and admission (Treatment period 1) to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the physician investigator, are acceptable. The presence of Left Bundle Branch Block (LBBB), atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Healthy on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel [excluding liver function tests], hematology [including coagulation], or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed/signed by the physician investigator
* Must be willing to adhere to the prohibitions and restrictions specified in this protocol
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* History of or current liver or renal insufficiency (estimated creatinine clearance below 60 milliliter per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the participant
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that, in the opinion of the investigator, with written concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* History of at least mild drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (latest edition DSM-5) criteria within 6 months before Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Plasma Concentration (Tmax) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  The Tmax is defined as actual sampling time to reach maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Relative Bioavailability of JNJ-54175446 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 hour post dose
  Relative bioavailability, calculated as individual Cmax and AUC treatment ratios (for the comparison of capsule to suspension formulation).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Baseline up to 9 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States